CLINICAL TRIAL: NCT02064842
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of TMC647055 in Combination With a Pharmacokinetic Enhancer (Part 1) Followed by an Open-label, Randomized, 3-way Crossover Study to Evaluate Short-term Safety, Tolerability and Pharmacokinetics of the Coadministration of TMC435, TMC647055 and a Pharmacokinetic Enhancer, at Steady-state (Part 2) in Healthy Japanese Subjects.
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of TMC647055 in Combination With Ritonavir (Part 1) and the Co-administration of TMC435, TMC647055 and Ritonavir (Part 2) in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR103540; TMC435HPC1011 (Other: Janssen R&D Ireland); 2013-004236-30 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy; TMC647055; TMC435; Simeprevir; Sovriad; Ritonavir (RTV)
MeSH Terms: interventions — 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione; Simeprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- TMC647055 150 mg or placebo + ritonavir (RTV) (Experimental): Participants in Part 1 will receive a single oral dose of 150 mg of TMC647055 or placebo with 30 mg of RTV on Day 1.
  Interventions: Drug: TMC647055; Drug: Placebo; Drug: Ritonavir (RTV)
- TMC647055 450 mg or placebo + RTV (Experimental): Participants in Part 1 will receive a single oral dose of 450 mg of TMC647055 or placebo with 30 mg of RTV on Day 1.
  Interventions: Drug: TMC647055; Drug: Placebo; Drug: Ritonavir (RTV)
- TMC647055 600 mg or placebo + RTV (Experimental): Participants in Part 1 will receive a single oral dose of 600 mg of TMC647055 or placebo with 30 mg of RTV on Day 1.
  Interventions: Drug: TMC647055; Drug: Placebo; Drug: Ritonavir (RTV)
- Sequence 1 (Treatment A-B-C) (Experimental): Participants in Part 2 will receive Treatment ABC in the following sequence - Treatment A: TMC435 150 mg once daily on Days 1 to 7; Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; and Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)
- Sequence 2 (Treatment B-C-A) (Experimental): Participants in Part 2 will receive Treatment BCA in the following sequence - Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; and Treatment A: TMC435 150 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)
- Sequence 3 (Treatment C-A-B) (Experimental): Participants in Part 2 will receive Treatment CAB in the following sequence - Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; Treatment A: TMC435 150 mg once daily on Days 1 to 7; and Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)
- Sequence 4 (Treatment A-C-B) (Experimental): Participants in Part 2 will receive Treatment ACB in the following sequence - Treatment A: TMC435 150 mg once daily on Days 1 to 7; Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; and Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)
- Sequence 5 (Treatment B-A-C) (Experimental): Participants in Part 2 will receive Treatment BAC in the following sequence - Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; Treatment A: TMC435 150 mg once daily on Days 1 to 7; and Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)
- Sequence 6 (Treatment C-B-A) (Experimental): Participants in Part 2 will receive Treatment CBA in the following sequence - Treatment C: TMC435 100 mg once daily + TMC647055 600 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; Treatment B: TMC435 75 mg once daily + TMC647055 450 mg once daily in combination with RTV 30 mg once daily on Days 1 to 7; and Treatment A: TMC435 150 mg once daily on Days 1 to 7 with a washout period of 7 days between consecutive treatment sessions in each individual participant.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir (RTV)

INTERVENTIONS:
Drug: TMC647055 — TMC647055 150 mg (1 capsule), 450 mg (3 capsules), 600 mg (4 capsules) taken orally (by mouth) once daily on Day 1 in Part 1. TMC647055 450 mg (3 capsules), and 600 mg (4 capsules) taken orally once daily on Days 1 to 7 in Part 2
Drug: TMC435 — TMC435 1 capsule of 75 mg, 100 mg, and 150 mg taken orally on Days 1 to 7 in Part 2
  Arms: Sequence 1 (Treatment A-B-C); Sequence 2 (Treatment B-C-A); Sequence 3 (Treatment C-A-B); Sequence 4 (Treatment A-C-B); Sequence 5 (Treatment B-A-C); Sequence 6 (Treatment C-B-A)
Drug: Placebo — Placebo capsule once daily taken orally on Day 1 in Part 1
  Arms: TMC647055 150 mg or placebo + ritonavir (RTV); TMC647055 450 mg or placebo + RTV; TMC647055 600 mg or placebo + RTV
Drug: Ritonavir (RTV) — RTV 30 mg (ie, 0.38 mL oral solution of RTV [80 mg/mL strength]) taken orally on Day 1 in Part 1 and on Days 1 to 7 in Part 2

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, and pharmacokinetics of TMC647055 in combination with ritonavir (Part 1); potential pharmacokinetic drug-drug interactions between TMC435 and the combination of TMC647055 with ritonavir; and to evaluate the short-term safety and tolerability when TMC435, TMC647055 and Ritonavir are co-administered (Part 2) in healthy Japanese participants.

DETAILED DESCRIPTION:
This is a single-center study which consists of 2 parts, sequentially conducted in 2 separate panels of 24 healthy adult Japanese participants each. Part 1 is a double-blinded (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (placebo is compared with the study medication to test whether the study medication has a real effect in clinical study), randomized (the study medication is assigned by chance) single ascending dose (SAD) part which will consist of a screening phase, a treatment phase, and a follow-up visit. Part 1 will have 3 cohorts (Cohort A, B, and C) with 8 participants each and they will be randomly assigned to receive either a single oral dose of TMC647055 (6 participants) or placebo (2 participants) in combination with RTV. The study duration for each participant will be approximately 5 weeks from screening to follow-up visit as maximum in Part 1. Part 2 is an open-label, randomized, 3-way crossover part which will consist of a screening phase, 3 treatment phases, and a follow-up phase. Each of the 24 participants will receive Treatment A, B, and C in 6 sequences (Treatment ABC, BCA, CAB, ACB, BAC, and CBA) with a washout period of at least 7 days between consecutive treatments. Safety evaluation will include assessment of adverse events, clinical laboratory tests, vital signs, electrocardiogram, and physical examination. The study duration for each participant will be approximately 10 weeks from screening to follow-up visit as maximum.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of Japanese descent who has resided outside Japan for no more than 5 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Must have signed an informed consent form
* Women must be of non-child-bearing potential (postmenopausal for at least 2 years, surgically sterile, or otherwise incapable of becoming pregnant)
* Women, except for postmenopausal women, should have a negative serum b-human chorionic gonadotropin pregnancy test at screening
* Men heterosexually active with a woman of childbearing potential must agree to use two effective methods of birth control, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study medication
* Must have a body mass index between 16.0 and 30.0 kg/m2, inclusive, and body weight not less than 45 kg at screening

Exclusion Criteria:

* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use within the past 1 year which in the Investigator's opinion would compromise participant's safety and/or compliance with the study procedures
* Participant's with Hepatitis A, B, or C infection, or human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2) infection at study screening
* Female participants who are breastfeeding at screening
* History of liver or renal impairment, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* History of clinically relevant skin disease or history of allergy to any medication

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with adverse events following the administration of TMC647055 | Up to Day 8
  Assessment will be following single oral doses of TMC647055/Ritonavir 150/30 mg, 450/30 mg and 600/30 mg
Part 1: Maximum observed plasma concentration of TMC647055 | Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose); Day 2 (24 and 36 hours postdose); Day 3; and in case of early withdrawal (once between Day 6 to 8)
  Assessment will be following single oral doses of TMC647055/Ritonavir 150/30 mg, 450/30 mg and 600/30 mg
Part 1: The actual sampling time to reach the maximum observed plasma of TMC647055 | Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose); Day 2 (24 and 36 hours postdose); Day 3; and in case of early withdrawal (once between Day 6 to 8)
  Assessment will be following single oral doses of TMC647055/Ritonavir 150/30 mg, 450/30 mg and 600/30 mg
Part 1: The actual sampling time of last measurable plasma concentration of TMC647055 | Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose); Day 2 (24 and 36 hours postdose); Day 3; and in case of early withdrawal (once between Day 6 to 8)
  Assessment will be following single oral doses of TMC647055/Ritonavir 150/30 mg, 450/30 mg and 600/30 mg
Part 1: Area under curve (AUC) of TMC647055 | Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose); Day 2 (24 and 36 hours postdose); Day 3; and in case of early withdrawal (once between Day 6 to 8)
  AUC from time 0 up to 24 hours after dosing, from time 0 to the time of the last measurable concentration, and from time 0 to infinite time will be assessed. Assessment will be following single oral doses of TMC647055/Ritonavir 150/30 mg, 450/30 mg and 600/30 mg
Part 2: Maximum observed plasma concentration of TMC435 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following TMC435 75 mg co-administered with TMC647055/ritonavir 450/30 mg; TMC435 100 mg co-administered with TMC647055/ritonavir 600/30 mg; and TMC435 150 mg alone
Part 2: The actual sampling time to reach the maximum observed plasma of TMC435 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following TMC435 75 mg co-administered with TMC647055/ritonavir 450/30 mg; TMC435 100 mg co-administered with TMC647055/ritonavir 600/30 mg; and TMC435 150 mg alone
Part 2: Area under curve (AUC) of TMC435 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  AUC from time 0 up to 24 hours after dosing will be assessed. Assessment will be following TMC435 75 mg co-administered with TMC647055/ritonavir 450/30 mg; TMC435 100 mg co-administered with TMC647055/ritonavir 600/30 mg; and TMC435 150 mg alone
Part 2: Maximum observed plasma concentration of TMC647055 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following TMC647055 600 mg co-administered with TMC435 100 mg and ritonavir 30 mg; and TMC647055 450 mg co-administered with TMC435 75 mg and ritonavir 30 mg
Part 2: The actual sampling time to reach the maximum observed plasma of TMC647055 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following TMC647055 600 mg co-administered with TMC435 100 mg and ritonavir 30 mg; and TMC647055 450 mg co-administered with TMC435 75 mg and ritonavir 30 mg
Part 2: Area under curve (AUC) of TMC647055 | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  AUC from time 0 up to 24 hours after dosing will be assessed. Assessment will be following TMC647055 600 mg co-administered with TMC435 100 mg and ritonavir 30 mg; and TMC647055 450 mg co-administered with TMC435 75 mg and ritonavir 30 mg

SECONDARY OUTCOMES:
Part 2: Maximum observed plasma concentration of ritonavir (RTV) | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following RTV 30 mg co-administered with TMC435 75 mg and TMC647055 450 mg; and RTV 30 mg co-administered with TMC435 100 mg and TMC647055 600 mg
Part 2: The actual sampling time to reach the maximum observed plasma of ritonavir (RTV) | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  Assessment will be following RTV 30 mg co-administered with TMC435 75 mg and TMC647055 450 mg; and RTV 30 mg co-administered with TMC435 100 mg and TMC647055 600 mg
Part 2: Area under curve (AUC) of ritonavir (RTV) | Day 1 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 2; Day 5; Day 6; Day 7 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose); Day 8; Day 9; Day 10; and end of treatment period or early withdrawal (once between Day 12 to 14)
  AUC from time 0 up to 24 hours after dosing will be assessed. Assessment will be following RTV 30 mg co-administered with TMC435 75 mg and TMC647055 450 mg; and RTV 30 mg co-administered with TMC435 100 mg and TMC647055 600 mg
Part 2: Number of participants with adverse events following the administration of TMC435 | Up to Day 14
  Assessment will be following TMC435 75 mg co-administered with TMC647055/ritonavir 450/30 mg; TMC435 100 mg co-administered with TMC647055/ritonavir 600/30 mg; and TMC435 150 mg alone

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Harrow, United Kingdom